CLINICAL TRIAL: NCT06961396
Title: Impact of Virtual Reality Combined With Manual Diaphragmatic Release on Adolescent Female With Painful Menstruation
Brief Title: Impact of Virtual Reality on Painful Menstruation
Acronym: VR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New Ismailia National University (Other)
Responsible Party: Principal Investigator, Mohamed Abdel Moeim Abo EL Ros, Assistant Professor of Pediatric Physical Therapy, New Ismailia National University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB # 21/3/20242025; IRB # 21/3/20242025 (Other: Zaytona University in Jordon)
Record Dates: First submitted 2025-04-08; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Painful Menstruation; Relaxation; Back Ligaments
Keywords: virtual reality; Diaphragmatic Releasing Technique; Painful Menstruation; Adolescent Female
MeSH Terms: conditions — Dysmenorrhea | interventions — Relaxation Therapy; Pain Management; Analgesia

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Who Masked: Participant
Masking Description: Using Sealed Envelopes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- virtual reality combined with diaphragmatic breathing technique (Experimental): to investigate the effect of virtual reality combined with the diaphragmatic breathing technique on painful menstruation, applied for 10 days successive 3 months
  Interventions: Device: Relaxation Technique; Device: Pain treatment
- cold LASER combined with diaphragmatic breathing technique (Experimental): to investigate the effect of cold LASER combined with diaphragmatic breathing technique on painful menstruation applied for 10 days successive 3 months
  Interventions: Device: Relaxation Technique; Device: Pain treatment

INTERVENTIONS:
Device: Relaxation Technique — utilizing virtual reality and a relaxation technique called diaphragmatic release to treat menstrual pain sufferers
  Other Names: Pain management
Device: Pain treatment — utilizing cold laser and a relaxation technique called diaphragmatic release to treat menstrual pain sufferers
  Other Names: Pain management

SUMMARY:
To investigate the effect of virtual reality on painful menstruation in adolescent female

DETAILED DESCRIPTION:
The focus of relatively recent work has been on non-pharmacological pain management techniques. The usage of virtual reality (VR) devices that can replicate three-dimensional (3D) immersive worlds is one particularly exciting advancement. This technology is becoming more widely available in healthcare settings and has shown promise in lowering pain and anxiety levels for people receiving minor gynecological disorders, dental work, burn wound care, and labor. So, the research purpose is targeted to look into the impact of virtual reality combined with diaphragmatic release as an active relaxation technique on painful menstruation in adolescent female

ELIGIBILITY:
Inclusion Criteria:

* age from 16 to 22 year
* cases of primary dysmenorrhea
* Normal body mass index (20-25)

Exclusion Criteria:

* cases with polycystic ovarian syndrome
* Obese female or body mass index more than 25
* severe bleeding with menstruation
* cases with low back pain due to orthopedic origin like disc herniation or spinal malalignment

Ages: 13 Years to 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — undergraduate students
Enrollment: 200 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
pain intensity | 1o days for successive three months
  Measurement of pain intensity using a visual analogue scale via the application of a virtual reality device combined with diaphragmatic release exercises

SECONDARY OUTCOMES:
Menstrual Distress Questionnaire | 1o days for successive three months
  detects the type and severity and type of symptoms of different changes even it is physical, , behavioral mood changes, and arousal symptoms during the different phases of the menstrual cycle

CONTACTS AND LOCATIONS:
Overall Officials: Hadeel MA Badwan, Ph.D, Study Chair — Al Zaytona University in Jordon
Locations (2):
- Mohamed Abdel Moenem Abo El Ros, Ismailia, Egypt
- Zaytona University in Jordon, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No
online sharing